CLINICAL TRIAL: NCT01018654
Title: Efficacy of Group Treatment for Hispanic Adolescents - RCT
Brief Title: Validating Interventions for Diverse Adolescents
Acronym: VIDA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00041220; K23DA019914 (NIH); 5K23DA19914-5
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2013-04

CONDITIONS: Substance-Related Disorders
Keywords: Substance Abuse; Substance Addiction
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Culturally Adapted Cognitive-Behavioral Treatment (Experimental): Culturally Adapted CBT for Substance Abuse
  Interventions: Behavioral: Culturally Adapted Cognitive-Behavioral Treatment
- Standard Cognitive-Behavioral Treatment (Active Comparator): Standard Cognitive-Behavioral Treatment for Substance Abuse
  Interventions: Behavioral: Standard Cognitive Behavioral Treatment

INTERVENTIONS:
Behavioral: Standard Cognitive Behavioral Treatment — Standard CBT for Substance Abuse
  Arms: Standard Cognitive-Behavioral Treatment
Behavioral: Culturally Adapted Cognitive-Behavioral Treatment — Culturally Adapted CBT for Substance Abuse
  Arms: Culturally Adapted Cognitive-Behavioral Treatment

SUMMARY:
The purpose of this study is to compare a culturally adapted and a non-culturally adapted group-based substance abuse treatment with Latino adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent between 13-18 years of age
* Parental consent
* Adolescent speaks English and Spanish
* Adolescent assent to participate in treatment and assessments
* Adolescent meets either DSM-IV diagnostic criteria for substance abuse or dependence
* Adolescent identifies as Hispanic

Exclusion Criteria:

* Adolescent younger than 13 or older than 18 years of age
* Adolescent requires higher level of care than what is provided in study
* Adolescent speaks only English or Spanish
* Parental consent not obtainable
* Adolescent does not assent to study
* Adolescent is overtly psychotic, severely depressed/suicidal, and/or presents with other mental disorder that will limit participation in group treatment
* Adolescent has completed substance abuse treatment elsewhere in the past 90 days
* Adolescent does not identify as Hispanic

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2010-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Substance Use Levels | Posttreatment, 3, 6, 12-month follow-ups

SECONDARY OUTCOMES:
Satisfaction with Treatment | Posttreatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States